CLINICAL TRIAL: NCT03001817
Title: A Phase 3, Multi-Center, Placebo-Controlled, Randomized, Double-Blind, 12-Week Study With a 40-Week, Active-Controlled, Double-Blind Extension to Evaluate the Efficacy and Safety of K-877 in Adult Patients With Fasting Triglyceride Levels ≥500 mg/dL and <2000 mg/dL and Normal Renal Function
Brief Title: Study to Evaluate the Efficacy and Safety of K-877 in Adult Patients With Fasting High Triglyceride Levels and Normal Renal Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K-877-301
Record Dates: First submitted 2016-11-29; First posted 2016-12-23 (Estimated); Results first posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Severe Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — K-877 compound; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 12 Week Efficacy (Placebo Comparator): K-877 or placebo comparator twice daily for 12 weeks
  Interventions: Drug: K-877; Drug: Placebo (for K-877)
- 40 Week Extension (Active Comparator): K-877 with placebo matching fenofibrate or fenofibrate with placebo matching K-877 for 40 weeks
  Interventions: Drug: K-877; Drug: Fenofibrate; Drug: Placebo (for K-877); Drug: Placebo (for Fenofibrate)

INTERVENTIONS:
Drug: K-877
Drug: Fenofibrate
  Arms: 40 Week Extension
Drug: Placebo (for K-877)
Drug: Placebo (for Fenofibrate)
  Arms: 40 Week Extension

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of K-877 in adult patients with fasting high triglyceride levels ≥500 mg/dL and <2000 mg/dL and normal renal function.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to comply with all study requirements and procedures throughout the duration of the study and give written informed consent;
2. Aged ≥18 years;
3. Patients receiving moderate- or high-intensity statin therapy must meet one of the following criteria¹ unless they have any exceptional conditions (see inclusion criterion 4):

   1. Aged ≥21 years with clinical atherosclerotic cardiovascular disease (ASCVD) (history of acute coronary syndrome or myocardial infarction, stable or unstable angina, coronary or other arterial revascularization, stroke, transient ischemic attack (TIA) presumed to be of atherosclerotic origin, or peripheral arterial disease or revascularization), on a high-intensity statin (or moderate-intensity statin if not a candidate for high-intensity statin due to safety concerns);
   2. Aged ≥21 years with a history of LDL-C ≥190 mg/dL, which is not due to secondary modifiable causes, on a high-intensity statin (or moderate-intensity statin if not a candidate for high-intensity statin due to safety concerns);
   3. Aged 40 to 75 years, inclusive, without clinical ASCVD but with diabetes and a history of LDL-C of 70 to 189 mg/dL, inclusive, on a moderate- or high-intensity statin; or
   4. Aged 40 to 75 years, inclusive, without clinical ASCVD or diabetes, with a history of LDL-C of 70 to 189 mg/dL, inclusive, with estimated 10-year risk for ASCVD of ≥7.5% by the Pooled Cohort Equation on a moderate- or high-intensity statin;
4. Patients currently on a low-intensity statin or not on a statin, must meet one of the following criteria:

   1. Patient does not meet any criteria for moderate- or high-intensity statin therapy listed above (see inclusion criteria, criterion 3.a. through 3.d.);
   2. Patient does meet one or more criteria for moderate- or high-intensity statin therapy listed above (see inclusion criteria 3.a. through 3.d.); but the patient is not a candidate for moderate or high-intensity statin due to safety concerns, or due to partial or complete statin intolerance; or
   3. Patient does meet one or more criteria for moderate- or high intensity statin therapy listed above (see inclusion criteria 3.b. through 3.d., except for 3.a.); but the patient is not a candidate for moderate or high-intensity statin for primary prevention after considering individual risk evaluation (e.g. current LDL C ≤70mg/dL) and patient preference;

Exclusion Criteria:

1. Patients who will require lipid-altering treatments other than study drugs (K-877 or fenofibrate), statins, ezetimibe, or PCSK9 inhibitors during the course of the study. These include bile acid sequestrants, non-study fibrates, niacin (>100 mg/day), omega-3 fatty acids (>1000 mg/day), or any supplements used to alter lipid metabolism including, but not limited to, red rice yeast supplements, garlic supplements, soy isoflavone supplements, sterol/stanol products, or policosanols;
2. Body mass index (BMI) >45 kg/m2 at Visit 1 (Week -8 or Week -6);
3. Patients with type 1 diabetes mellitus;
4. Patients with newly diagnosed (within 3 months prior to Visit 2 [Week -2]) or poorly controlled type 2 diabetes mellitus (T2DM), defined as hemoglobin A1c >9.5% at Visit 1 (Week -8 or Week -6);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (220):
- United States (110):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Cahaba Research, Inc., Birmingham, Alabama
  - Boyett Health Services Inc, Hamilton, Alabama
  - Longwood Research - Saadat Ansari, MD, LLC, Huntsville, Alabama
  - Terence T. Hart, MD, Tuscumbia, Alabama
  - Arrowhead Health Centers, Glendale, Arizona
  - Phoenix Medical Research Institute, LLC, Peoria, Arizona
  - Elite Clinical Studies, Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - iResearch - Little Rock, Little Rock, Arkansas
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Advanced Research Center, Anaheim, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - Downtown L.A. Research Center, Inc., Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Lucita M. Cruz, MD., Inc., Norwalk, California
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - Atlantic Clinical Research Collaborative, Boynton Beach, Florida
  - ALL Medical Research, LLC, Cooper City, Florida
  - S & W Clinical Research, Fort Lauderdale, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - AMPM Research Clinic, Miami Gardens, Florida
  - Advanced Research Institute Inc, New Port Richey, Florida
  - Ocala Cardiovascular Research, Ocala, Florida
  - South Florida Research Solutions LLC. - Pembroke Pines, Pembroke Pines, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Meridien Research - Tampa, Tampa, Florida
  - Columbus Regional Health, Columbus, Georgia
  - Physicians Research Associates, Inc, Lawrenceville, Georgia
  - Georgia Institute for Clinical Research, Marietta, Georgia
  - Meridian Clinical Research - Savannah, GA, Savannah, Georgia
  - Solaris Clinical Research, Meridian, Idaho
  - Apex Medical Research - Illinois, Chicago, Illinois
  - Lemah Creek Clinical Research, Melrose Park, Illinois
  - Koch Family Medicine, Morton, Illinois
  - Community Hospital of Anderson and Madison County, Inc, Anderson, Indiana
  - American Health Network - Avon Clinical Research Department, Avon, Indiana
  - Medisphere Medical Research Center, Evansville, Indiana
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - The Iowa Clinic - Cardiovascular Services, West Des Moines, Iowa
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Research Integrity LLC, Owensboro, Kentucky
  - Clinical Trials Management, LLC - Northshore, Covington, Louisiana
  - Clinical Trials Management LLC - Southshore, Metairie, Louisiana
  - Clinical Trials of America, LLC - West Monroe, LA, West Monroe, Louisiana
  - Maryland Cardiovascular Specialist, Baltimore, Maryland
  - Aa Mrc, Llc, Flint, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - David M. Headley, MD P.A., Port Gibson, Mississippi
  - Consult and Research Associates, St Louis, Missouri
  - Advance Clinical Research, Inc, St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Desert Endocrinology Clinical Research Center - Henderson, Henderson, Nevada
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Lakeshore Primary Care Associate, Hamburg, New York
  - Mid-Hudson Medical Research, PLLC - Hopewell Junction, New Windsor, New York
  - Mid-Hudson Medical Research, PLLC - New Windsor, New Windsor, New York
  - Orchard Park Family Practice, Orchard Park, New York
  - Diabetes and Endocrinology Consultants, P.C., Morehead City, North Carolina
  - Lillestol Research, LLC, Fargo, North Dakota
  - Sterling Research Group, Ltd. - Auburn, Cincinnati, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Alpha Research Associates, LLC, Dayton, Ohio
  - Prestige Clinical Research, Franklin, Ohio
  - Ohio Clinical Research - Lyndhurst, Lyndhurst, Ohio
  - Rama Research LLC, Marion, Ohio
  - RAS Health Ltd, Marion, Ohio
  - Summit Research Group, LLC, Munroe Falls, Ohio
  - Ohio Clinical Research, LLC - Willoughby Hills, Willoughby Hills, Ohio
  - South Oklahoma Heart Research, Oklahoma City, Oklahoma
  - Clinical Research Associates of Central PA, LLC, Altoona, Pennsylvania
  - Harleysville Medical Associates, Harleysville, Pennsylvania
  - Richard M.Kastelic MD and Associates, Johnstown, Pennsylvania
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Center for Medical Research, LLC, Providence, Rhode Island
  - DeGarmo Institute Of Medical Research, Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - PMG Research of Bristol, LLC - State, Bristol, Tennessee
  - New Phase Research & Development - Knoxville, Knoxville, Tennessee
  - Clinical Research Solutions - Smyrna, TN, Smyrna, Tennessee
  - Health Innovation Research Group, Arlington, Texas
  - DCT-AACT, LLC, dba Discovery Clinical Trials, Austin, Texas
  - Inquest Clinical Research, Baytown, Texas
  - Protenium Clinical Research, LLC - Dallas, Dallas, Texas
  - VA North Texas Health Care System - Dallas VA Medical Center (DVAMC), Dallas, Texas
  - Academy of Diabetes, Thyroid and Endocrine, P.A., El Paso, Texas
  - Juno Research, LLC - Northwest Site, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Juno Research, LLC - Southwest Houston Site, Houston, Texas
  - Pioneer Research Solutions Inc., Houston, Texas
  - Grace Research, LLC - Huntsville, TX, Huntsville, Texas
  - Protenium Clinical Research, LLC, Hurst, Texas
  - Juno Research, LLC - Katy, Katy, Texas
  - FMC Science, Lampasas, Texas
  - DCT - McAllen Primary Care, LLC, McAllen, Texas
  - San Antonio Premier Internal Medicine, San Antonio, Texas
  - Physician PrimeCare Research Institute, PLLC dba Health Texas Research Institute, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Bandera Family HealthCare Research, LLC (BFHC), San Antonio, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - York Clinical Research LLC, Norfolk, Virginia
  - Exemplar Research Inc. - Fairmont, WV, Morgantown, West Virginia
  - Allegiance Research Specialists, LLC, Wauwatosa, Wisconsin
- Belarus (10):
  - Brest Regional Hospital, Brest
  - Grodno University Hospital, Grodno
  - Gomel Regional Clinical Center of Cardiology, Homyel
  - Gomel Regional Clinical Hospital, Homyel
  - City Clinical Hospital #10, Minsk
  - City Clinical Hospital #1, Minsk
  - Minsk Regional Clinical Hospital, Minsk
  - Minsk Scientific and Practice Center of Surgery, Transplantology and Hematology, Minsk
  - Mogilev Regional Medical and Diagnostic Center, Mogilev
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Bulgaria (9):
  - Medical Center Diamedical 2013 OOD, Dimitrovgrad
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski EAD- First Cardiology Clinic, Pleven
  - University Multiprofile Hospital for Active Treatment Dr. Georgi Stranski EAD- Second Cardiology Clinic, Pleven
  - UMHAT Sveti Georgi - Clinic of Cardiology, Plovdiv
  - MHAT Dr. Bratan Shukjerov, Smolyan
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD, Smolyan
  - Fifth Multiprofile Hospital for Active Treatment - Sofia EAD - Department of Cardiology, Sofia
  - Fifth Multiprofile Hospital for Active Treatment - Sofia EAD - Department of Endocrinology and Meteorism Diseases, Sofia
  - Medical Center Orfey OOD, Stara Zagora
- Czechia (8):
  - Lipidova poradna, Bílina
  - Medicus Services SRO, Brandýs nad Labem
  - Fakultni nemocnice Hradec Kralove, Klinika gerontologicka a metabolicka, Hradec Králové
  - Onkologicka klinika 2. LF UK a FN Motol, Prague
  - Ordinace pro choroby srdce a cev, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Oblastni nemocnice Trutnov, Oddeleni klinicke biochemie, Trutnov
  - MUDr. Nina Zemkova s.r.o. Interni Ambulance, Uherské Hradište
- Georgia (8):
  - Unimed Ajara LLC, Batumi
  - Clinic LJ Ltd, Kutaisi
  - Aleksandre Aladashvili Clinic - LLC, Tbilisi
  - Archangel St Michael Multiprofile Clinical Hospital Ltd, Tbilisi
  - Emergency Cardiology Center by Academician G. Chapidze Ltd, Tbilisi
  - Institute of Clinical Cardiology Ltd, Tbilisi
  - Unimed Kakheti - Caraps Medline LLC, Tbilisi
  - Unimed Kakheti - Telavi Referral Hospital LLC, Telavi
- Hungary (9):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - DRC Balatongyorok, Balatongyörök
  - Dr Lakatos Ferenc Belgyogyaszati-Kardiologiai Maganrendelo, Békéscsaba
  - Magyar Honvedseg Allami Egeszsegugyi Kozpont, II. sz Belgyogyaszat Osztaly, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - BKS Research Kft., Hatvan
  - Pecsi Tudomanyegyetem Klinikai Kozpont I.sz. Belgyogyaszati Klinika, Pécs
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Poland (12):
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Kardiologii, lek. med. Krzysztof Cymerman, Gdynia
  - SALVIA Lekston i Madej s.j., Katowice
  - Malopolskie Centrum Alergii i Immunoterapii Allmedis SP Z O O, Krakow
  - AppleTreeClinics Sp. z o.o., Lodz
  - NZOZ All - Med Centrum Medyczne Specjalistyczne Gabinety Lekarskie Marcin Ogorek, Lodz
  - Nzoz Salusmed, Lodz
  - MEDICOME Sp. z o.o., Oświęcim
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne OMEGA SP Z O O, Płock
  - Clinmedica Research Omc Sp z o.o. Sp, Skierniewice
  - Centrum Kardiologiczne Pro Corde Sp. z o. o., Wroclaw
- Russia (41):
  - City Clinical Hospital n.a. M.P. Konchalovskiy, Zelenograd, Moscow
  - First City Clinical Hospital n.a. E.E.Volosevich, Arkhangelsk
  - Northern Medical Clinical Center named after N.A. Semashko of the Federal Medical and Biological Agency, Arkhangelsk
  - Altay Regional Cardiology Dispensary, Cardiology Department for Patients with Acute Myocardial Infarction, Barnaul
  - Chita State Medical Academy, Chita
  - Interregional Clinical Diagnostic Center, Kazan'
  - Kazan State Medical University based at City Clinical Hospital #7, Kazan'
  - Federal State Budget Institution "Scientific-Research Institute of Complex Problems of Cardiovascular Diseases", Kemerovo
  - Medical Center "Alliance", Kirovsk
  - Krasnoyarsk State Medical University n.a. prof. V.F. Voino-Yasenetsky, Krasnoyarsk
  - Central Clinical Hospital of Russian Academy of Sciences, Moscow
  - City Clinical Hospital #15 n.a. O.M. Filatov, Moscow
  - City Clinical Hospital n.a. M.E. Zhadkevich of Moscow Healthcare Department, Moscow
  - Federal State Budget Institution "Outpatient Clinic #3" of Russian Federation President's Management Department, Moscow
  - National Medical Research Center of Cardiology - Department of Atherosclerosis, Moscow
  - National Medical Research Center of Cardiology, Moscow
  - National Medical Research Center of Preventive Medicine, Moscow
  - Non-governmental Private Healthcare Institution "Scientific Clinical Centre of Open Joint-Stock Company Russian Railways" (JSC "RZD"), Moscow
  - City Clinical Hospital No.2, Novosibirsk
  - RC Medical LLC, Novosibirsk
  - Research Institute of Physiology and Fundamental Medicine, Novosibirsk
  - Orenburg State Medical University based at City Clinical Hospital #1, Orenburg
  - Clinical-diagnostic center "Zdorovye", Rostov-on-Don
  - Rostov-on-Don City Hospital of Emergency Care, Rostov-on-Don
  - Almazov National Medical Research Centre, Scientific Laboratory of Electrocardiology, Saint Petersburg
  - Almazov National Medical Research Centre, Saint Petersburg
  - BioTechService LLC, Saint Petersburg
  - City hospital #38 n.a. N.A. Semashko, Saint Petersburg
  - Clinic Complex JSC, Saint Petersburg
  - Clinical Hospital #122 n. a. L.G. Sokolov of the Federal Medical Biological Agency, Saint Petersburg
  - Consultative Diagnostic Center with Out-patient Clinic, Saint Petersburg
  - Limited Liability Company "MedPomosch", Saint Petersburg
  - Medical Technologies LLC, Saint Petersburg
  - North-Western State Medical University named after I.I. Mechnikov, Saint Petersburg
  - Saint-Petersburg State Budget Healthcare Institution "City Pokrovskaya Hospital", Cardiology Departmen, Saint Petersburg
  - Regional Clinical Cardiology Dispensary, Saratov
  - Saratov State Medical University n. a. V.I. Razumovsky, Saratov
  - Tomsk National Research Medical Center of Russian Academy of Sciences, Tomsk
  - Autonomous Institution of healthcare of the Voronezh region "Voronezh regional clinical consultative and diagnostic centre, Voronezh
  - Yaroslavl Regional Clinical Hospital for War Veterans - International Center on the Problems of the Elderly "Zdorovoe Dolgoletie", Yaroslavl
  - Ural State Medical University based at Central City Clinical Hospital No.1 of Oktyabrskiy District, Yekaterinburg
- Ukraine (13):
  - Ivano-Frankivsk Regional Clinical Cardiological Dispensary, Chronic Ischaemic Heart Disease Department, Ivano-Frankivsk
  - JSC "Ukrainian Railways" Kharkiv Railway Clinical Hospital#1 of Branch "Healthcare Center" of PJSC "Ukrainian Railways", Cardiology Depart #1, Kharkiv
  - JSC "Ukrainian Railways" Kharkiv Railway Clinical Hospital#1 of Branch "Healthcare Center" of PJSC "Ukrainian Railways", Cardiology Depart #2, Kharkiv
  - Municipal Non-Commercial Enterprise "City Clinical Emergency Hospital n.a. prof. O.I. Meshchaninov" of Kharkiv City Council, Kharkiv
  - Municipal Noncommercial Enterprise "City Clinical Hospital #27" of Kharkiv City Council, Kharkiv
  - Municipal Noncommercial Enterprise "City Outpatient Clinic #9" of Kharkiv City Council, Kharkiv
  - Kyiv City Clinical Hospital #1, Urgent Cardiology Department, Kyiv
  - Limited Liability Company "Treatment and Diagnostic Center "Adonis Plus"", Outpatient Department, Kyiv
  - SI "Institute of Gerontology n.a. D.F.Chebotarev NAMS of Ukraine", Cardiol. Un. of Clin. Physiology and Int. Organs Path. Dep-t., Gen. Ther.Unit, Kyiv
  - SI "Institute of Gerontology n.a. D.F.Chebotarev NAMS of Ukraine", Cardiol. Un. of Clin. Physiology and Int. Organs Path. Dep-t, Kyiv
  - Municipal Institution "City Clinical Hospital #3 n.a. prof. L.J. Aleinikova", Cardiology Intensive Therapy Department, Odesa
  - Small Private Enterprise, Medical Centre "Puls", Vinnytsia
  - Municipal Institution "City Clinical Hospital #6", Therapeutic Department, Zaporizhzhia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible participants entered a 4- to 6-week lifestyle stabilization period followed by a 2-week TG qualifying period, used to determine eligibility for the study. After confirmation of qualifying fasting TG values, eligible participants entered a 12-week Efficacy Period. Participants who successfully completed the 12-week Efficacy Period were eligible to continue in a 40-week Extension Period.
Groups:
- K-877: Participants randomized to receive K-877 0.2 mg tablets twice daily in the 12-week Efficacy Period continued to receive K-877 0.2 mg tablets twice daily (BID) as well as placebo matching fenofibrate tablets once daily, in the 40-week Extension Period
- Placebo/Fenofibrate: Participants randomized to receive placebo matching K-877 0.2 mg tablets BID in the 12-week Efficacy Period received fenofibrate 145 mg tablet once daily and placebo matching K-877 0.2 mg tablet BID in the 40-week Extension Period.
Period: 12 Week Efficacy
Arm/Group | K-877 | Placebo/Fenofibrate
Started | 368 | 183
Completed (Including 2 participants (one participant each group) who skipped Week 12 but did not discontinue study drug and entered the 40-week Extension Period.) | 356 | 179
Not Completed | 12 | 4
Period: 40 Week Extension
Arm/Group | K-877 | Placebo/Fenofibrate
Started (Note that 8 participants (6 participants in the K-877 group and 2 participants in the placebo/fenofibrate 145 mg group) withdrew after completing the 12-week Efficacy Period and did not start the 40-week Extension Period.) | 350 | 177
Completed | 335 | 163
Not Completed | 15 | 14

BASELINE CHARACTERISTICS:
Groups:
- K-877: Participants randomized to receive K-877 0.2 mg BID in the 12-week Efficacy Period continued to receive K-877 0.2 mg BID, as well as placebo matching fenofibrate 145 mg once daily, in the 40-week Extension Period.
- Placebo/Fenofibrate: Participants randomized to receive placebo matching K-877 0.2 mg BID in the 12-week Efficacy Period received fenofibrate 145 mg once daily and placebo matching K-877 0.2 mg BID in the 40-week Extension Period.
- Total: Total of all reporting groups
Arm/Group | K-877 | Placebo/Fenofibrate | Total
Number analyzed (Participants) | 368 | 183 | 551
Age, Customized [Count of Participants; unit: Participants]
  Age (Years): <65 | 351 | 176 | 527
  Age (Years): ≥65 | 17 | 7 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 39 | 136
  Male | 271 | 144 | 415
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 8 | 35
  Not Hispanic or Latino | 341 | 175 | 516
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 4 | 0 | 4
  White | 358 | 180 | 538
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 810.98 (369.284) | 819.25 (414.722) | 813.73 (384.611)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Fasting Triglyceride(TG) Levels From Baseline to Week 12
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Groups:
- K-877: K-877 0.2 mg tablet BID
- Placebo: Placebo matching K-877 0.2 mg tablet BID
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent of Change | -56.00 [-72.08 to -32.40] | -7.97 [-44.78 to 49.87]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

2. Secondary Outcome: Percent Change From Baseline to Week 12 in Remnant Cholesterol
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -52.95 [-67.97 to -27.64] | -3.36 [-31.18 to 39.47]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

3. Secondary Outcome: Percent Change From Baseline to Week 12 in HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 16.25 [-1.13 to 40.15] | 4.00 [-8.91 to 15.58]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann Method

4. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo A1
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 1.21 [-8.68 to 11.77] | 2.13 [-5.75 to 9.48]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.5443, Hodges-Lehmann method

5. Secondary Outcome: Percent Change From Baseline to Week 12 in Non-HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -16.07 [-31.98 to 0.73] | 0.81 [-17.14 to 22.65]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann Method

6. Secondary Outcome: Percent Change From Baseline to Week 12 in Total Cholesterol
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -11.26 [-24.95 to 3.40] | 1.55 [-13.17 to 19.84]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

7. Secondary Outcome: Percent Change From Baseline to Week 12 in LDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 31.93 [0.84 to 78.12] | 1.01 [-19.83 to 26.41]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

8. Secondary Outcome: Percent Change From Baseline to Week 12 in Free Fatty Acids (FFAs)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Chage
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 356 | 171
Percent Chage | -19.07 [-41.64 to 14.10] | 10.29 [-22.61 to 71.16]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

9. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo A2
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 15.30 [0.32 to 27.06] | 2.89 [-5.99 to 9.71]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

10. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo B
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 2.41 [-12.71 to 19.36] | 3.73 [-9.09 to 17.51]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.4939, Hodges-Lehmann method

11. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo B48
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -31.35 [-64.59 to 33.65] | 22.62 [-38.27 to 138.37]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

12. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo B100
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 3.09 [-12.20 to 20.48] | 2.76 [-11.55 to 17.15]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.8371, Hodges-Lehmann method

13. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo C2
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 0.00 [-25.01 to 0.00] | 0.00 [-0.03 to 0.00]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.3415, Hodges-Lehmann method

14. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo C3
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -39.56 [-54.84 to -16.27] | 5.11 [-17.61 to 36.39]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

15. Secondary Outcome: Percent Change From Baseline to Week 12 in Apo E
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -28.48 [-43.33 to -3.58] | 0.56 [-18.21 to 37.20]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

16. Secondary Outcome: Change From Baseline to Week 12 in Fibroblast Growth Factor 21 (FGF21)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
pg/mL | 196.97 [37.42 to 469.14] | 3.88 [-100.26 to 121.23]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

17. Secondary Outcome: Change From Baseline to Week 12 in hsCRP
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
mg/L | -0.051 [-1.491 to 0.743] | -0.100 [-1.273 to 0.597]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.7442, Hodges-Lehmann method

18. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Very Low-Density Lipoprotein (VLDL) Cholesterol-Large
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -27.89 [-51.25 to -0.45] | 5.99 [-21.19 to 39.53]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

19. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Very Low-Density Lipoprotein (VLDL) Cholesterol-Intermediate
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -17.32 [-37.38 to 5.09] | 4.70 [-18.69 to 28.96]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

20. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Very Low-Density Lipoprotein (VLDL) Cholesterol-Small
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -4.13 [-19.85 to 16.25] | 1.86 [-18.40 to 24.46]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0374, Hodges-Lehmann method

21. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Intermediate Density Lipoproteins 1
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 4.47 [-13.54 to 24.49] | 2.10 [-17.05 to 25.95]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.7429, Hodges-Lehmann method

22. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Intermediate Density Lipoproteins 2
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 15.50 [-0.61 to 44.88] | 3.06 [-14.55 to 24.51]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

23. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins I
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 45.24 [11.80 to 87.52] | 1.04 [-15.53 to 21.64]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

24. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins IIa
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 59.36 [17.64 to 112.28] | 0.75 [-16.59 to 22.46]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

25. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins IIb
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 61.87 [12.77 to 111.62] | 1.26 [-17.93 to 26.00]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

26. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins IIIa
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 33.08 [-10.18 to 85.81] | 0.85 [-14.11 to 33.65]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

27. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins IIIb
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -1.50 [-41.65 to 52.99] | 1.11 [-19.55 to 29.73]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.3669, Hodges-Lehmann method

28. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins IVa
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -24.88 [-56.93 to 7.48] | -0.26 [-20.30 to 25.74]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

29. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins IVb
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -34.81 [-53.95 to -12.17] | 5.60 [-19.62 to 32.04]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

30. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Low Density Lipoproteins IVc
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -21.68 [-39.22 to -4.57] | 4.65 [-14.87 to 24.95]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

31. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - High Density Lipoproteins 2b
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -7.34 [-19.80 to 3.85] | 2.04 [-10.69 to 15.52]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

32. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - High Density Lipoproteins 3 and 2a
Description: Two lipoprotein subclasses, HDL3 and HDL2a, were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -2.01 [-13.44 to 9.82] | 1.76 [-9.43 to 11.91]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0509, Hodges-Lehmann method

33. Secondary Outcome: Percent Change From Baseline to Week 12 in Ion Mobility - Major LDL Particle Measurement
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 2.38 [0.74 to 4.31] | -0.06 [-0.97 to 0.84]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

34. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - VLDL & Chylomicron Particles
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | -37.93 [-60.09 to -7.54] | 5.37 [-23.57 to 53.56]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

35. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - VLDL & Chylomicron Particles-Large
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | -48.58 [-73.96 to -15.98] | 7.54 [-35.11 to 103.86]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

36. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - VLDL Particles-Medium
Time Frame: 12 Weeks
Population: Since there were one or multiple records with a baseline value of 0, the percent change cannot be determined for such records. In such cases, the secondary endpoints were evaluated for change from baseline to week 12.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
nmol/L | -33.57 [-72.83 to 0.59] | 7.58 [-33.08 to 47.63]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

37. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - VLDL Particles-Small
Time Frame: 12 Weeks
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
nmol/L | 0.90 [-13.53 to 18.10] | -1.87 [-23.39 to 12.26]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0647, Hodges-Lehmann method

38. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - LDL Particles (Total)
Time Frame: 12 Weeks
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
nmol/L | 209.41 [-139.84 to 596.86] | 51.43 [-213.52 to 275.68]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0007, Hodges-Lehmann method

39. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - Intermediate-density Lipoprotein (IDL) Particles
Time Frame: 12 Weeks
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
nmol/L | -5.52 [-109.19 to 49.33] | -0.21 [-98.28 to 102.41]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.1399, Hodges-Lehmann method

40. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - LDL Particles-Large
Time Frame: 12 Weeks
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
nmol/L | 27.54 [0.00 to 256.61] | 0.00 [0.00 to 39.76]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0122, Hodges-Lehmann method

41. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - LDL Particles-Small
Time Frame: 12 Weeks
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
nmol/L | 87.75 [-254.51 to 468.78] | 23.85 [-200.74 to 297.25]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0994, Hodges-Lehmann method

42. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - HDL Particles (Total)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | 2.87 [-9.72 to 17.11] | -1.07 [-12.86 to 13.72]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0904, Hodges-Lehmann method

43. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - HDL Particles-Large
Time Frame: 12 Weeks
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: μmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
μmol/L | 0.27 [-0.94 to 1.45] | 0.05 [-1.28 to 1.43]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.4346, non-parametric Hodges-Lehmann method

44. Secondary Outcome: Change From Baseline to Week 12 in Lipoprotein Fraction - HDL Particles-Medium
Time Frame: 12 Weeks
Population: as for outcome 36
Measure: Median (Inter-Quartile Range); unit: μmol/L
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
μmol/L | -0.97 [-4.31 to 2.65] | 0.02 [-3.32 to 2.74]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.1474, non-parametric Hodges-Lehmann method

45. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - HDL Particles-Small
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | 7.08 [-14.34 to 32.08] | -2.42 [-18.72 to 17.47]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0054, non-parametric Hodges-Lehmann method

46. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - VLDL Particle Size
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | -5.70 [-14.70 to 5.21] | 0.80 [-10.18 to 12.05]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0002, Hodges-Lehmann method

47. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - LDL Particle Size
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 364 | 180
Percent Change | 1.00 [0.00 to 3.26] | 0.01 [-0.51 to 1.00]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

48. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - HDL Particle Size
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | -1.14 [-4.44 to 2.07] | 0.00 [-2.89 to 3.36]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.0118, Hodges-Lehmann method

49. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - Triglyceride (Total)
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | -48.78 [-69.80 to -18.51] | 8.43 [-28.90 to 70.31]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

50. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - VLDL & Chylomicron Triglyceride
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 367 | 182
Percent Change | -49.06 [-70.30 to -20.13] | 6.71 [-28.59 to 70.18]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < .0001, Hodges-Lehmann method

51. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipoprotein Fraction - HDL Cholesterol
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 358 | 170
Percent Change | -0.11 [-19.62 to 22.54] | -4.63 [-18.43 to 13.68]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.2049, Hodges-Lehmann method

52. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of TG:HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -62.64 [-79.05 to -34.09] | -11.22 [-49.07 to 57.86]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

53. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of Total Cholesterol (TC):HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -25.84 [-42.29 to -4.77] | -3.86 [-22.83 to 19.87]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

54. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of Non-HDL-C:HDL-C
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -30.79 [-47.69 to -5.64] | -4.49 [-25.49 to 23.46]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

55. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of LDL-C:Apo B
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 30.90 [7.30 to 62.27] | -0.49 [-21.23 to 18.79]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

56. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of Apo B:Apo A1
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | 0.73 [-15.39 to 20.43] | 2.47 [-11.55 to 14.60]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p = 0.9117, Hodges-Lehmann method

57. Secondary Outcome: Percent Change From Baseline to Week 12 in Lipid and Lipoprotein Ratios of Apo C3:Apo C2
Time Frame: 12 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo
Number analyzed (Participants) | 368 | 183
Percent Change | -24.84 [-44.79 to -3.68] | 7.50 [-13.29 to 35.11]
Statistical Analysis 1: Comparison: K-877 vs Placebo; Test type: Superiority; p < 0.0001, Hodges-Lehmann method

58. Secondary Outcome: Percent Change From Baseline to Week 52 in Fasting TG
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 335 | 163
Percent of Change | -57.93 [-73.76 to -31.97] | -55.45 [-68.95 to -28.74]

59. Secondary Outcome: Percent Change From Baseline to Week 52 in Remnant Cholesterol
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 331 | 161
Percent of Change | -53.98 [-70.63 to -26.55] | -49.11 [-67.45 to -21.35]

60. Secondary Outcome: Percent Change From Baseline to Week 52 in HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 335 | 163
Percent of Change | 17.65 [-1.27 to 39.29] | 19.35 [3.03 to 38.89]

61. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo A1
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 334 | 162
Percent of Change | 1.63 [-8.59 to 10.42] | 3.48 [-3.42 to 10.92]

62. Secondary Outcome: Percent Change From Baseline to Week 52 in Non-HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 335 | 163
Percent of Change | -17.24 [-32.00 to 0.00] | -15.71 [-29.85 to 0.63]

63. Secondary Outcome: Percent Change From Baseline to Week 52 in TC
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 335 | 163
Percent of Change | -11.84 [-25.37 to 1.61] | -9.93 [-23.08 to 3.21]

64. Secondary Outcome: Percent Change From Baseline to Week 52 in LDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 331 | 161
Percent of Change | 31.15 [2.04 to 70.59] | 36.84 [1.38 to 78.29]

65. Secondary Outcome: Percent Change From Baseline to Week 52 in FFAs
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 263 | 128
Percent of Change | -18.08 [-40.81 to 18.60] | -13.64 [-38.15 to 13.91]

66. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo A2
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 333 | 162
Percent of Change | 9.26 [-2.44 to 22.58] | 12.31 [0.00 to 22.58]

67. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo B
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 334 | 162
Percent of Change | 0.93 [-12.65 to 19.85] | 2.46 [-12.68 to 17.00]

68. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo B48
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 333 | 161
Percent of Change | -14.04 [-56.90 to 68.32] | -5.22 [-48.40 to 84.46]

69. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo B100
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 333 | 161
Percent of Change | 1.48 [-13.93 to 19.77] | 1.97 [-12.66 to 17.23]

70. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo C2
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 330 | 159
Percent of Change | -8.70 [-30.60 to 0.00] | -1.80 [-24.20 to 0.00]

71. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo C3
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 160
Percent of Change | -36.70 [-58.82 to -15.25] | -30.77 [-51.65 to -5.91]

72. Secondary Outcome: Percent Change From Baseline to Week 52 in Apo E
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent of Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent of Change | -29.94 [-47.16 to -10.64] | -30.67 [-44.60 to -4.44]

73. Secondary Outcome: Change From Baseline to Week 52 in FGF21
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
pg/mL | 259.20 [16.10 to 545.65] | 207.50 [53.70 to 499.90]

74. Secondary Outcome: Change From Baseline to Week 52 in hsCRP
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 333 | 162
mg/L | 0.000 [-1.000 to 1.400] | -0.200 [-1.320 to 0.400]

75. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - VLDL Cholesterol-Large
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -33.43 [-53.96 to 5.54] | -24.44 [-46.64 to 4.31]

76. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - VLDL Cholesterol-Intermediate
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -21.71 [-40.18 to 11.94] | -11.70 [-32.94 to 10.50]

77. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - VLDL Cholesterol-Small
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -4.28 [-22.23 to 17.29] | -3.23 [-18.03 to 28.03]

78. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Intermediate Density Lipoproteins 1
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 4.44 [-12.86 to 25.81] | 8.23 [-15.88 to 37.67]

79. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Intermediate Density Lipoproteins 2
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 21.05 [2.32 to 48.91] | 21.09 [-4.00 to 51.00]

80. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins I
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 48.52 [17.51 to 95.70] | 38.99 [9.07 to 82.58]

81. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins IIa
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 64.54 [21.24 to 120.44] | 44.52 [8.87 to 113.47]

82. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins IIb
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 58.07 [14.25 to 122.86] | 42.18 [8.41 to 102.42]

83. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins IIIa
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 31.63 [-7.19 to 75.36] | 30.84 [-3.26 to 86.03]

84. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins IIIb
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 0.34 [-42.86 to 42.90] | 4.31 [-23.03 to 45.81]

85. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins IVa
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -24.86 [-55.96 to 10.11] | -15.38 [-48.48 to 13.31]

86. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins IVb
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -35.58 [-52.93 to -11.22] | -27.86 [-50.00 to -2.41]

87. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Low Density Lipoproteins IVc
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -24.00 [-36.55 to -6.88] | -22.02 [-35.80 to -3.57]

88. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - High Density Lipoproteins 2b
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -9.54 [-18.19 to 2.06] | -8.99 [-19.00 to 1.5]

89. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - High Density Lipoproteins 3 and 2a
Description: Two lipoprotein subclasses, HDL3 and HDL2a, were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | -3.58 [-12.59 to 6.5] | -3.06 [-12.33 to 6.09]

90. Secondary Outcome: Percent Change From Baseline to Week 52 in Ion Mobility - Diameter of the Major LDL Particle
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 332 | 162
Percent Change | 2.38 [0.55 to 4.69] | 1.56 [0.39 to 3.37]

91. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - VLDL & Chylomicron Particles
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | -39.09 [-59.18 to -7.46] | -30.29 [-53.45 to 2.58]

92. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - VLDL & Chylomicron Particles-Large
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | -51.64 [-75.46 to -10.20] | -51.23 [-70.89 to 2.75]

93. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - VLDL Particles-Medium
Time Frame: 52 Weeks
Population: Since there were one or multiple records with a baseline value of 0, the percent change cannot be determined for such records. In such cases, the secondary endpoints were evaluated for change from baseline to week 52.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
nmol/L | -34.20 [-71.10 to -1.20] | -20.70 [-70.4 to 15.00]

94. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - VLDL Particles-Small
Time Frame: 52 Weeks
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
nmol/L | 0.00 [-19.00 to 19.40] | 3.85 [-21.90 to 21.80]

95. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - LDL Particles (Total)
Time Frame: 52 Weeks
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
nmol/L | 193.00 [-115.00 to 533.00] | 213.50 [-97.00 to 572.00]

96. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - IDL Particles
Time Frame: 52 Weeks
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
nmol/L | -9.00 [-101.00 to 48.00] | -6.50 [-133.00 to 75.00]

97. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - LDL Particles-Large
Time Frame: 52 Weeks
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
nmol/L | 25.50 [0.00 to 280.00] | 50.50 [0.00 to 215.00]

98. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - LDL Particles-Small
Time Frame: 52 Weeks
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
nmol/L | 81.00 [-222.00 to 420.00] | 138.00 [-187.00 to 436.00]

99. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - HDL Particles
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | 1.07 [-11.50 to 15.46] | 1.38 [-12.57 to 12.45]

100. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - HDL Particles-Large
Time Frame: 52 Weeks
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
umol/L | 0.10 [-1.20 to 1.40] | -0.10 [-1.20 to 1.20]

101. Secondary Outcome: Change From Baseline to Week 52 in Lipoprotein Fraction - HDL Particles-Medium
Time Frame: 52 Weeks
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: umol/L
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
umol/L | -0.80 [-4.80 to 2.10] | -1.15 [-4.10 to 2.00]

102. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - HDL Particles-Small
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | 9.01 [-11.19 to 32.20] | 6.37 [-12.50 to 30.46]

103. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - VLDL Particle Size
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | -6.12 [-16.22 to 5.41] | -6.70 [-16.08 to 5.51]

104. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - LDL Particle Size
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 286 | 143
Percent Change | 0.99 [0.00 to 3.08] | 0.51 [0.00 to 2.54]

105. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - HDL Particle Size
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | -1.15 [-4.49 to 2.33] | -1.11 [-3.49 to 2.33]

106. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - Triglyceride
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | -48.01 [-70.62 to -22.77] | -48.29 [-65.74 to -7.86]

107. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - VLDL & Chylomicron Triglyceride
Description: Two types of lipoprotein particles were analyzed together as one measurement without distinction.
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 302 | 150
Percent Change | -48.38 [-71.40 to -24.22] | -47.69 [-65.55 to -7.72]

108. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipoprotein Fraction - HDL Cholesterol
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 256 | 121
Percent Change | -3.88 [-18.74 to 22.40] | -2.63 [-17.24 to 12.90]

109. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of TG:HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 335 | 163
Percent Change | -63.46 [-80.92 to -32.83] | -65.21 [-77.40 to -38.31]

110. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of TC:HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 335 | 163
Percent Change | -27.21 [-42.91 to -6.46] | -27.59 [-41.20 to -6.65]

111. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of Non-HDL-C:HDL-C
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 335 | 163
Percent Change | -30.63 [-48.39 to -7.52] | -32.36 [-46.88 to -8.11]

112. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of LDL-C:Apo B
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 326 | 157
Percent Change | 28.03 [6.73 to 57.69] | 24.73 [2.50 to 60.32]

113. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of Apo B:Apo A1
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 334 | 162
Percent Change | 1.05 [-16.67 to 18.46] | -1.76 [-13.04 to 14.58]

114. Secondary Outcome: Percent Change From Baseline to Week 52 in Lipid and Lipoprotein Ratios of Apo C3:Apo C2
Time Frame: 52 Weeks
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | K-877 | Placebo/Fenofibrate
Number analyzed (Participants) | 329 | 159
Percent Change | -20.98 [-40.38 to -0.74] | -13.99 [-37.76 to 6.76]

ADVERSE EVENTS:
Time Frame: 52 Weeks
Description: Treatment-emergent adverse event (TEAE) was defined as any adverse event that occurred for the first time after the first dose of double-blind study drug or existed prior to the first dose and worsened during the post-dosing period.
Groups:
- K-877: 12-Week Efficacy: * K-877 0.2 mg Tablets BID
  * Only AEs with onset in the 12-week efficacy period are included.
- Placebo: 12-Week Efficacy: * Placebo matching K-877 0.2 mg BID
  * Only AEs with onset in the 12-week efficacy period are included.
- K-877 and Fenofibrate Placebo: 40-Week Extension: * Participants randomized to receive K-877 0.2 mg tablets twice daily in the 12-week Efficacy Period continued to receive K-877 0.2 mg tablets BID, as well as placebo matching fenofibrate 145 mg tablets once daily, in the 40-week Extension Period.
  * Only AEs with onset in the 40-week extension period are included.
- Fenofibrate and K-877 Placebo: 40-Week Extension: * Participants randomized to receive placebo matching K-877 0.2 mg tablets BID in the 12-week Efficacy Period received fenofibrate 145 mg tablets once daily and placebo matching K-877 0.2 mg tablets BID in the 40-week Extension Period.
  * Only AEs with onset in the 40-week extension period are included.
Arm/Group | K-877: 12-Week Efficacy | Placebo: 12-Week Efficacy | K-877 and Fenofibrate Placebo: 40-Week Extension | Fenofibrate and K-877 Placebo: 40-Week Extension
All-Cause Mortality (participants affected / at risk) | 0/368 | 0/183 | 3/350 | 0/177
Serious Adverse Events (participants affected / at risk) | 13/368 | 5/183 | 17/350 | 3/177
Other Adverse Events (participants affected / at risk) | 3/368 | 2/183 | 9/350 | 9/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | K-877: 12-Week Efficacy (N=368) | Placebo: 12-Week Efficacy (N=183) | K-877 and Fenofibrate Placebo: 40-Week Extension (N=350) | Fenofibrate and K-877 Placebo: 40-Week Extension (N=177)
Angina unstable (Cardiac disorders) | 2 | 1 | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 1 | 0 | 0
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Allergic granulomatous angiitis (Immune system disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
Glomerulonephritis chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral artery aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-877: 12-Week Efficacy (N=368) | Placebo: 12-Week Efficacy (N=183) | K-877 and Fenofibrate Placebo: 40-Week Extension (N=350) | Fenofibrate and K-877 Placebo: 40-Week Extension (N=177)
Nasopharyngitis (Infections and infestations) | 3 | 2 | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (5):
  • Study Protocol: ver.1.0 (2016-09-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03001817/Prot_000.pdf
  • Study Protocol: ver.2.0 (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT03001817/Prot_001.pdf
  • Statistical Analysis Plan: v1.0 (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT03001817/SAP_002.pdf
  • Statistical Analysis Plan: v2.0 (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03001817/SAP_003.pdf
  • Statistical Analysis Plan: Addendum (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT03001817/SAP_004.pdf